CLINICAL TRIAL: NCT06014970
Title: The Health and Wellness Curriculum Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Victor Carrion (Other)
Collaborators: Pure Edge Inc. (Unknown); University of San Diego (Other); University of South Carolina (Other); Iowa State University (Other)
Responsible Party: Sponsor-Investigator, Victor Carrion, Professor and Vice-Chair of Psychiatry and Behavioral Sciences, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-31715
Record Dates: First submitted 2023-08-13; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Trauma, Psychological; Stress, Psychological
MeSH Terms: conditions — Psychological Trauma; Stress, Psychological | interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health and Wellness Curriculum (Experimental): Trained instructors will provide the Health and Wellness Curriculum at the Ravenswood City schools. Each school receiving the curriculum will have a dedicated space and receive a 30 minute class twice a week. Through group discussion, nutrition and character education, and breathing exercises, students will receive instruction to focus their attention, calm their minds, reduce stress, and think before reacting.
  Interventions: Behavioral: Health and Wellness Curriculum
- Control (No Intervention): All control participants go through the same assessment procedures as the experimental group without any intervention.

INTERVENTIONS:
Behavioral: Health and Wellness Curriculum — The curriculum includes instructions, activities, and lessons on mindfulness, neurobiology, meditation, positive thinking, movement, and nutrition.
  Arms: Health and Wellness Curriculum

SUMMARY:
The overarching goal of the study is to examine the effects of a new Health and Wellness Curriculum (Pure Power) being implemented in the Ravenswood City School District in East Palo Alto. The Pure Power Curriculum, which the Sonima Foundation (Now Pure Edge Inc.,)developed, includes exercise based on yoga, common exercise regimes, relaxation techniques, mindfulness practices, and nutrition education, and was introduced in 2014 to the Ravenswood City Schools, independent of the research. The new curriculum was expected to yield dramatic positive effects on students' socio-emotional development, which the investigators aimed to examine through this study.

This research evaluation measures the impact of the Pure Power Curriculum on the socioemotional, behavioral, cognitive, academic, and physiological functioning of students in a low-socioeconomic status (SES) school community over time by evaluating student development at three time points: baseline (i.e., prior to implementation of the curriculum), one-year follow-up, and two-year follow-up. Only third and fifth-grade students were eligible for enrollment at baseline. All data collection procedures were replicated with the control group.

DETAILED DESCRIPTION:
Participants for the experimental group were recruited from the Ravenswood City School District.

Trained instructors provided the Health and Wellness Curriculum at the Ravenswood City schools. Each school receiving the curriculum had a dedicated space and received a 30-minute class twice a week. Through group discussion, nutrition and character education, and breathing exercises, students received instruction to focus their attention, calm their minds, reduce stress, and think before reacting.

Control subjects were recruited from Orchard School District, Alum Rock Union Elementary School District, and nearby community organizations/ after-school programs (like Boys and Girls Clubs) in the San Francisco Bay Area. The control group was recruited after the experimental group had finished baseline data collection.

At three separate points over the course of three years, all consenting participants received academic and neurobehavioral assessments via paper questionnaires in the classroom. The research staff measured children's academic functioning abilities and moods, thoughts, and behavioral symptoms, which were employed as a control variable in the proposed analyses. This was accomplished by administering the Wide Range Achievement Test (WRAT IV), the Behavior Assessment System for Children (BASC-II), the Responses to Stress Questionnaire, and the Behavior Rating Inventory of Executive Function (BRIEF).

At Ravenswood, at least 100 students from the original 800-student sample were recruited for the cognitive (plus additional questionnaires), sleep, and endocrinology portions of the study. From this 100-student sub-sample, at least 30 students were recruited to participate in the neuroimaging component of the study. Cognitive abilities were assessed using the Kaufman Assessment Battery for Children 2 (K-ABC II): all scales and subtests. During the cognitive testing portion of the study, participants also completed the reading section of the Wide Range Achievement Test (WRAT-IV) and the Trauma Symptoms Checklist for Children (TSCC).

This project was the first systematic neuroscience study of skill-building in children via a multi-method assessment that includes structural MRI, functional MRI, salivary cortisol, and sleep architecture data. These are methods that have proven critical in the fundamental understanding of stress in children. The research will identify critical biopsychosocial components responsible for cognitive, behavioral, emotional, and academic improvement, effective implementation, and the sustainability of the program.

Diurnal salivary cortisol was collected by parents using the Salimetrics Children's Swab for 2 consecutive days at five specific times: within 20 minutes of waking up, before breakfast, before lunch, before dinner and before bedtime. Results from these time periods will serve as an index of baseline cortisol rhythmicity. This process occurred a total of three times (once at each assessment time).

fMRI: Children completed the Tanner stages form to assess their scale of physical development (puberty) and handedness form to determine if they are right or left-handed and the Domain-Specific Impulsivity Scale for Children (DSIS-C) questionnaire, which measures impulsivity traits in the domains of schoolwork and interpersonal relationships, to be used in concert with neuroimaging data. fMRI, DTI and sMRI data will be acquired on a 3T scanner with a state-of-the-art 32-channel parallel imaging coil. Children will perform up to four cognitive and emotional experiments during fMRI scanning:

* A stop signal task investigated brain plasticity in systems associated with attention and cognitive control.
* An emotional labeling task was used to examine brain plasticity in systems associated with emotion perception.

Data for each experiment was acquired across 2 runs (except only 1 run for the emotional labeling task), each lasting 6 minutes, in order to minimize fatigue while providing adequate statistical power to detect effects of interest. This process will occur a total of three times (once at each assessment time). Participants will also complete a Delay Discounting Task outside of the MRI scanner.

Two salivary cortisol samples were collected by researchers: one at the beginning of the scan and the other one after the scan. One salivary hormone sample was collected at the end of the scan.

To assess sleep, researchers conducted the overnight ambulatory polysomnography (PSG) of sleep.

ELIGIBILITY:
Inclusion Criteria:

* All 3rd and 5th-grade students in the participating school districts

Exclusion Criteria:

* For fMRI:

  1. History of trauma involving head injury.
  2. Metal in or on the body that cannot be removed(braces, piercings or tattoos).
  3. Consistent exposure to metal(i.e. hobbies grinding metal).
  4. Pregnancy.
  5. Left-handedness.
  6. Any tattoos on the body, including eyeliner and other permanent makeup.
* For general study: Students who demonstrate the inability to follow all study procedures during a specific assessment will be excluded from that portion of the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1176 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Mean Change in Response to Stress Questionnaire | Three time points: Baseline, 12 months, 24 months
  The Response to Stress Questionnaire (RSQ) is comprised of a checklist of stressors that may be experienced during stressful situations. Following the checklist of stressors, a possible total of 57 questions ask individuals how they respond to stressors they recently experienced. Youth rate how often they cope with a stressor in a certain way on a 4-point Likert scale (ranging from 1, "Not at all," to 4, "A lot"). The RSQ is divided into two major subscales: School-Related Stress Experiences and Stress Reactivity. Stress Reactivity is further divided into two composite scores: involuntary engagement and primary control. To score the RSQ, proportion scores are created for each factor to control for individual differences in rates of endorsing items. Changes in scores will be assessed between all time points.
Mean Change in School Achievement | Three time points: Baseline, 12 months, 24 months
  School achievement was assessed with the Wide Range Achievement Test-Revised Spelling and Math scale score. The spelling subscale was a phonetic test that assessed the degree to which students could encode sounds into written words. The math computation subscale measured students' ability to identify numbers, count, and solve written computational problems. The scores are summed across the subscales and scaled according to the standardized score. A higher score reflects a higher performance. Changes in scores will be assessed between all time points.
Mean Change in Emotional and Behavioral Dysregulation | Three time points: Baseline, 12 months, 24 months
  Internalizing symptoms (i.e. anxiety and depression) and externalizing problems (i.e. attention and hyperactivity) were assessed via a self-report version of the Behavior Assessment System for Children, 2nd edition (BASC-II). For items 1-69, participants were asked to respond True or False to a series of statements about themselves. For items 70-176 participants were asked to respond Never, Sometimes, Often, or Almost Always to a series of statements about themselves. Responses were scored via the BASC-II formulas for subscale t-scores, percentiles, and validity scores. Changes in scores will be assessed between all time points.
Change from Baseline of Diurnal Salivary Cortisol | Three time points: Baseline, 12 months, 24 months
  Diurnal salivary cortisol were collected by parents using the Salimetrics Children's Swab for 2 consecutive days at five specific times. Results from these time periods will serve as an index of baseline cortisol rhythmicity. This process will occur a total of three times (once at each assessment time).
Change from Baseline of Sleep Quality | Three time points: Baseline, 12 months, 24 months
  Research staff employed the Compumedics Safiroambulatory Polysomnography monitoring system to assess sleep. This ambulatory device includes a cap and several electrodes, and records electroencephalogram (EEG), Electromyography (EMG), expiratory/inspiratory nasal airway pressure, nasal/oral airflow, finger pulse oximetry, electrocardiogram (ECG), movements of the rib cage and abdomen, snoring, body position and bilateral anterior tibialis EMG.
Change from Baseline of Sleep Habits | Three time points: Baseline, 12 months, 24 months
  Parents complete the abbreviated Child's Sleep Habits Questionnaire (CSHQ). Parents are asked to recall sleep behaviors occurring over a "typical" recent week. Items are rated on a three-point scale: "usually" if the sleep behavior occurred five to seven times/week; "sometimes" for two to four times/week; and "rarely" for zero to one time/week. Some items were reversed in order to consistently make a higher score indicative of more disturbed sleep. This process will occur a total of three times (once at each assessment time).
Measure of Brain Plasticity for Attention and Cognitive Control | Three time points: Baseline, 12 months, 24 months
  fMRI task: A stop signal task was used to investigate brain plasticity in systems associated with attention and cognitive control. In stop signal task, participants made button presses in response to left/right-pointing arrows and occasionally cancel their prepared responses. Data for each experiment will be acquired across 2 runs (except only 1 run for the emotional labeling task), each lasting 6 minutes, in order to minimize fatigue while providing adequate statistical power to detect effects of interest. This process will occur a total of three times (once at each assessment time).
Measure of Brain Plasticity for Risk Taking and Risk Avoidance | Three time points: Baseline, 12 months, 24 months
  fMRI task: A balloon analogue risk task (BART) will be used to investigate brain plasticity in systems associated with risk-taking and risk avoidance. In BART, participants choose between pumping a balloon or to cash out on each trial. Every successful pump adds to their reward on that trial. If the balloon explodes, the accumulated earning on that trial will be lost.
Measure of Brain Plasticity for Emotion Perception | Three time points: Baseline, 12 months, 24 months
  fMRI task: Participants will decide which of two facial expressions presented on the bottom of the screen match the facial expression at the top of the screen. The faces have either angry or fearful expression.
Measure of Brain Plasticity for Emotional Control | Three time points: Baseline, 12 months, 24 months
  fMRI task: Participants viewed 60 neutral and aversive images which are carefully selected for pediatric populations based on previous studies. When participants see the instructional cue "Look", participants naturally react to the picture. When participants see the cue "Decrease", participants tell themselves a story about the picture to feel less negative (i.e., to reappraise). Prior to the fMRI experiment, children will be given examples about how to reappraise (e.g., imagining it is just a scene from a movie) and asked to report the reappraisals aloud during training to ensure understanding of the instructions.

SECONDARY OUTCOMES:
Overall Cognitive Assessment | Three time points: Baseline, 12 months, 24 months
  Cognitive abilities were assessed using the Kaufman Assessment Battery for Children 2 (K-ABCII): all scales and subtests. Scores are summed across the subtests and higher scores reflect higher performance on each scale.